CLINICAL TRIAL: NCT03342300
Title: Comparing the Effectiveness and Toxicity for Locally Advanced, Unresectable or Metastatic Soft-tissue Sarcoma Patients Who Had Received Total Dose of Anthracycline Antibiotics More Than 300mg/m2 With Pegylated Liposomal Doxorubicin Versus Pirarubicin Plus Ifosfamide, Dacarbazine, a Multicentre, Open-label, Randomised Phase 2 Trial
Brief Title: Pegylated Liposomal Doxorubicin Versus Pirarubicin Plus Ifosfamide, Dacarbazine in Locally Advanced, Unresectable or Metastatic Soft-tissue Sarcoma
Acronym: PDVPSTS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Chinese PLA General Hospital (Other); Beijing Jishuitan Hospital (Other); Xijing Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBTRA-03
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Progression-free Survival; Overall Survival; Toxicity
Keywords: soft tissue sarcoma; pegylated liposomal doxorubicin; pirarubicin; toxicity for heart; cumulative dose
MeSH Terms: conditions — Sarcoma | interventions — liposomal doxorubicin; pirarubicin

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (1:1) to receive pegylated liposomal doxorubicin (50 mg/m² on day 1 of every 21-day cycle for up to six cycles) or pirarubicin (60 mg/m² on day 1 of every 21-day cycle for up to six cycles) plus ifosfamide (2 g/m²/d d2-4 of every 21-day cycle for up to six cycles) and dacarbazine (300 mg/m²/d d2-4 of every 21-day cycle for up to six cycles).
Who Masked: Outcomes Assessor
Masking Description: A web-based central randomisation with block sizes of two and four was stratified by extent of disease,anthracycline administration method, and previous systemic therapy. Participants and investigators will not be masked to treatment assignment. The primary endpoint will be assessed in the intention-to-treat population. The outcome assessors will be masked to the two research groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): participants will recieve pegylated liposomal doxorubicin (50 mg/m²d1) plus ifosfamide (2 g/m²/d d2-3), dacarbazine (300 mg/m²/d d2-3).
  Interventions: Drug: pegylated liposomal doxorubicin
- Arm B (Placebo Comparator): participants will recieve pirarubicin (60 mg/m²d1) plus ifosfamide (2 g/m²/d d2-3), dacarbazine (300 mg/m²/d d2-3).
  Interventions: Drug: pirarubicin

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin — Several efforts have been made to improve the toxicity profile of conventional anthracyclines, including the use of liposomal encapsulation technology,such as pegylated liposomal doxorubicin.
  Arms: Arm A
Drug: pirarubicin — Another effort has been made to improve the toxicity profile of conventional anthracyclines is the development of novel anthracycline analogs,such as pirarubicin.
  Arms: Arm B

SUMMARY:
Advanced soft tissue sarcoma patients who have previously recieved anthracyclines might still benefit from doxorubicin, ifosfamide and dacarbazine. However doxorubicin might be stopped using because of chronic cumulative heart toxicity. Several efforts have been made to improve the toxicity profile of conventional anthracyclines, including the use of liposomal encapsulation technology and the development of novel anthracycline analogs,such as pegylated liposomal doxorubicin and pirarubicin. However their actual effectiveness and toxicity have not been studied in prospective trial. The purpose of the study is to investigate whether they are available for this group of patients.

DETAILED DESCRIPTION:
We design this multicentre, open-label, randomised, phase 2 trial at 5 academic hospitals in China. Eligible patients need to be aged 16 years or older with a diagnosis of an advanced unresectable or metastatic soft-tissue sarcoma, of intermediate or high grade, for which no standard curative therapy will be available, an Eastern Cooperative Oncology Group performance status of 0-1, and measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1.

Participants will be randomly assigned (1:1) to receive pegylated liposomal doxorubicin (60 mg/m² via continuous intravenous infusion for 4-6 h on day 1 of every 21-day cycle for up to six cycles) or pirarubicin (30 mg/m2/d continuous intravenous infusion for 3h on day 1 and 2 of every 21-day cycle for up to six cycles) plus ifosfamide ( 2 g/m²/d intravenously for 2h on day 2,3 and 4 of every 21-day cycle for up to six cycles), dacarbazine (300 mg/m²/d intravenously for 2h on day 2,3 and 4 of every 21-day cycle for up to six cycles ).After six cycles of treatment, patients will be followed up expectantly whereas patients with stable or responsive disease are allowed to continue with ifosfamide and dacarbzine until documented disease progression. A web-based central randomisation with block sizes of two and four was stratified by extent of disease, drug administration method, and previous systemic therapy. Patients and investigators will not be masked to treatment assignment. The primary endpoint is progression survival, analysed in the intention-to-treat population. Safety analyses will be done in all patients who receive any amount of study drug.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older;
* diagnosis of an advanced unresectable or metastatic soft tissue sarcoma, of intermediate or high grade, for which no standard curative therapy is available;
* cumulative dose of anthracycline antibiotic ≥ 300mg/m2;
* stable or responsive to doxorubicin, potential beneficiary;
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, a life expectancy of at least 3 months;
* measurable disease according to RECIST 1.1;
* adequate end-organ and haemopoietic function.

Exclusion Criteria:

* progress over doxorubicin;
* previous mediastinal or cardiac radiotherapy;
* a low-grade tumour according to standard grading systems (eg, American Joint Committee on Cancer grade 1 and 2 or Fédération Nationale des Centres de Lutte Contre le Cancer grade 1);
* significant cardiac dysfunction;
* severe chronic obstructive pulmonary disease;
* a known infection with HIV or active infection with hepatitis B or hepatitis C;
* known brain metastases unless previously treated and well controlled for a period of 3 months or longer;
* combination with other anti-tumor therapy;
* pregnant or breastfeeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 12 weeks
  Progression-free survival is defined as time from randomisation to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment or randomisation.

SECONDARY OUTCOMES:
overall survival | 12 months
  overall survival is defined as the duration from date of randomisation to the date of death from any cause.
objective response rate, ORR | 12 weeks
  objective response rate includes complete and partial responses as defined by RECIST version 1.1.
left ventricular ejection fraction function | 12 months
  We use ultrasound to routinely estimate the left ventricular ejection fraction function.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D.and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, CSR

REFERENCES:
- [Background] Frezza AM, Stacchiotti S, Gronchi A. Systemic treatment in advanced soft tissue sarcoma: what is standard, what is new. BMC Med. 2017 Jun 2;15(1):109. doi: 10.1186/s12916-017-0872-y. PMID 28571564
- [Background] Antman K, Crowley J, Balcerzak SP, Rivkin SE, Weiss GR, Elias A, Natale RB, Cooper RM, Barlogie B, Trump DL, et al. An intergroup phase III randomized study of doxorubicin and dacarbazine with or without ifosfamide and mesna in advanced soft tissue and bone sarcomas. J Clin Oncol. 1993 Jul;11(7):1276-85. doi: 10.1200/JCO.1993.11.7.1276. PMID 8315425
- [Background] Jelic S, Kovcin V, Milanovic N, Babovic N, Kreacic M, Ristovic Z, Vlajic M, Filipovic-Ljeskovic I. Randomised study of high-dose epirubicin versus high-dose epirubicin-cisplatin chemotherapy for advanced soft tissue sarcoma. Eur J Cancer. 1997 Feb;33(2):220-5. doi: 10.1016/s0959-8049(96)00297-3. PMID 9135492
- [Background] Le Cesne A, Judson I, Crowther D, Rodenhuis S, Keizer HJ, Van Hoesel Q, Blay JY, Frisch J, Van Glabbeke M, Hermans C, Van Oosterom A, Tursz T, Verweij J. Randomized phase III study comparing conventional-dose doxorubicin plus ifosfamide versus high-dose doxorubicin plus ifosfamide plus recombinant human granulocyte-macrophage colony-stimulating factor in advanced soft tissue sarcomas: A trial of the European Organization for Research and Treatment of Cancer/Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 2000 Jul;18(14):2676-84. doi: 10.1200/JCO.2000.18.14.2676. PMID 10894866
- [Background] Santoro A, Tursz T, Mouridsen H, Verweij J, Steward W, Somers R, Buesa J, Casali P, Spooner D, Rankin E, et al. Doxorubicin versus CYVADIC versus doxorubicin plus ifosfamide in first-line treatment of advanced soft tissue sarcomas: a randomized study of the European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 1995 Jul;13(7):1537-45. doi: 10.1200/JCO.1995.13.7.1537. PMID 7602342
- [Background] Tap WD, Jones RL, Van Tine BA, Chmielowski B, Elias AD, Adkins D, Agulnik M, Cooney MM, Livingston MB, Pennock G, Hameed MR, Shah GD, Qin A, Shahir A, Cronier DM, Ilaria R Jr, Conti I, Cosaert J, Schwartz GK. Olaratumab and doxorubicin versus doxorubicin alone for treatment of soft-tissue sarcoma: an open-label phase 1b and randomised phase 2 trial. Lancet. 2016 Jul 30;388(10043):488-97. doi: 10.1016/S0140-6736(16)30587-6. Epub 2016 Jun 9. PMID 27291997
- [Background] Bui-Nguyen B, Butrynski JE, Penel N, Blay JY, Isambert N, Milhem M, Kerst JM, Reyners AK, Litiere S, Marreaud S, Collin F, van der Graaf WT; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group (EORTC/STBSG) and the Sarcoma Alliance for Research through Collaboration (SARC). A phase IIb multicentre study comparing the efficacy of trabectedin to doxorubicin in patients with advanced or metastatic untreated soft tissue sarcoma: the TRUSTS trial. Eur J Cancer. 2015 Jul;51(10):1312-20. doi: 10.1016/j.ejca.2015.03.023. Epub 2015 Apr 23. PMID 25912752
- [Background] Schoffski P, Ray-Coquard IL, Cioffi A, Bui NB, Bauer S, Hartmann JT, Krarup-Hansen A, Grunwald V, Sciot R, Dumez H, Blay JY, Le Cesne A, Wanders J, Hayward C, Marreaud S, Ouali M, Hohenberger P; European Organisation for Research and Treatment of Cancer (EORTC) Soft Tissue and Bone Sarcoma Group (STBSG). Activity of eribulin mesylate in patients with soft-tissue sarcoma: a phase 2 study in four independent histological subtypes. Lancet Oncol. 2011 Oct;12(11):1045-52. doi: 10.1016/S1470-2045(11)70230-3. Epub 2011 Sep 19. PMID 21937277
- [Background] Lefrak EA, Pitha J, Rosenheim S, Gottlieb JA. A clinicopathologic analysis of adriamycin cardiotoxicity. Cancer. 1973 Aug;32(2):302-14. doi: 10.1002/1097-0142(197308)32:23.0.co;2-2. No abstract available. PMID 4353012
- [Background] Vondrakova D, Malek F, Ostadal P, Vranova J, Miroslav P, Schejbalova M, Neuzil P. Correlation of NT-proBNP, proANP and novel biomarkers: copeptin and proadrenomedullin with LVEF and NYHA in patients with ischemic CHF, non-ischemic CHF and arterial hypertension. Int J Cardiol. 2011 Aug 4;150(3):343-4. doi: 10.1016/j.ijcard.2011.05.029. Epub 2011 Jun 2. No abstract available. PMID 21640398
- [Background] Von Hoff DD, Layard MW, Basa P, Davis HL Jr, Von Hoff AL, Rozencweig M, Muggia FM. Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med. 1979 Nov;91(5):710-7. doi: 10.7326/0003-4819-91-5-710. PMID 496103
- [Background] Rivankar S. An overview of doxorubicin formulations in cancer therapy. J Cancer Res Ther. 2014 Oct-Dec;10(4):853-8. doi: 10.4103/0973-1482.139267. PMID 25579518
- [Background] Nielsen OS, Dombernowsky P, Mouridsen H, Daugaard S, Van Glabbeke M, Kirkpatrick A, Verweij J. Epirubicin is not Superior to Doxorubicin in the Treatment of Advanced Soft Tissue Sarcomas.The Experience of the EORTC Soft Tissue and Bone Sarcoma Group. Sarcoma. 2000;4(1-2):31-5. doi: 10.1155/S1357714X00000062. PMID 18521432
- [Background] Judson I, Radford JA, Harris M, Blay JY, van Hoesel Q, le Cesne A, van Oosterom AT, Clemons MJ, Kamby C, Hermans C, Whittaker J, Donato di Paola E, Verweij J, Nielsen S. Randomised phase II trial of pegylated liposomal doxorubicin (DOXIL/CAELYX) versus doxorubicin in the treatment of advanced or metastatic soft tissue sarcoma: a study by the EORTC Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2001 May;37(7):870-7. doi: 10.1016/s0959-8049(01)00050-8. PMID 11313175
- [Background] Bafaloukos D, Papadimitriou C, Linardou H, Aravantinos G, Papakostas P, Skarlos D, Kosmidis P, Fountzilas G, Gogas H, Kalofonos C, Dimopoulos AM. Combination of pegylated liposomal doxorubicin (PLD) and paclitaxel in patients with advanced soft tissue sarcoma: a phase II study of the Hellenic Cooperative Oncology Group. Br J Cancer. 2004 Nov 1;91(9):1639-44. doi: 10.1038/sj.bjc.6602148. PMID 15494721
- [Background] Poveda A, Lopez-Pousa A, Martin J, Del Muro JG, Bernabe R, Casado A, Balana C, Sanmartin O, Menendez MD, Escudero P, Cruz J, Belyakova E, Menendez D, Buesa JM. Phase II Clinical Trial With Pegylated Liposomal Doxorubicin (CAELYX(R)/Doxil(R)) and Quality of Life Evaluation (EORTC QLQ-C30) in Adult Patients With Advanced Soft Tissue Sarcomas: A study of the Spanish Group for Research in Sarcomas (GEIS). Sarcoma. 2005;9(3-4):127-32. doi: 10.1080/13577140500287024. PMID 18521419
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347